CLINICAL TRIAL: NCT06203977
Title: Inflammation REduction to Prevent cArdiovascular Injury in Renal Disease (REPAIR)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Hamilton Academic Health Sciences Organization (Other); St. Joseph's Health Care London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REPAIR
Record Dates: First submitted 2023-12-08; First posted 2024-01-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases; Renal Failure
Keywords: Tolerance; Colchicine Resistance; Hematologic markers
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Phase 1 basket trial including 2 open-label single-arm cohorts: REPAIR CKD cohort and REPAIR Dialysis cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- REPAIR CKD cohort (Active Comparator): Patients will receive open label colchicine 0.3 mg daily for 8 weeks followed, in patients who tolerated the 0.3 mg dose, by forced titration to 0.6 mg daily for 8 weeks.
  Interventions: Drug: Colchicine
- REPAIR Dialysis cohort (Active Comparator): Patients will receive open label colchicine 0.3 mg daily for 8 weeks followed, in patients who tolerated the 0.3 mg dose, by forced titration to 0.6 mg daily for 8 weeks.
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — 0.3mg and 0.6mg tablets

SUMMARY:
Phase 1 basket trial including 2 open-label single-arm cohorts: REPAIR CKD cohort and REPAIR Dialysis cohort. Open label colchicine 0.3 mg daily for 8 weeks followed, in patients who tolerated the 0.3 mg dose, by forced titration to 0.6 mg daily for 8 weeks.

DETAILED DESCRIPTION:
The REPAIR CKD cohort will enroll 100 patients with chronic kidney disease not requiring dialysis. The REPAIR Dialysis cohort will enroll 100 patients with chronic kidney disease requiring chronic maintenance dialysis. Each participant will be followed for up to 17 weeks, to determine among adults with severe chronic kidney disease not requiring dialysis and (separately) in those requiring dialysis, the proportion who, over 8 weeks of treatment, discontinue colchicine 1) 0.3 mg daily and 2) 0.6 mg daily.

ELIGIBILITY:
Inclusion Criteria:

1. One of either:

   1.2 Estimated GFR using CKD-EPI 2021 equation of ≤30 ml/min/1.73m2 on at least two occasions separated by at least 2 months and do not yet require dialysis and are not expected by their treating nephrologist to require dialysis in the next 6 months (REPAIR CKD cohort), or 1.3 receiving chronic maintenance dialysis 2 or more times per week for the previous 90 days (REPAIR Dialysis cohort);
2. Age ≥18 years
3. Provide informed consent to participate.

Exclusion Criteria:

1. Currently treated with and cannot withdraw colchicine due to medical necessity; or
2. Known allergy/sensitivity to colchicine; or
3. Prior self-reported intolerance to colchicine at a dose of 0.6 mg daily or lower; or
4. Currently pregnant or planning to become pregnant or breastfeed during the study; or
5. Of childbearing potential AND do not have a negative pregnancy test OR do not agree to use two forms of contraception for the duration of the study; or
6. Anticipated living donor renal transplant within the next 6 months; or
7. Using a strong inhibitor of p-glycoprotein or strong inhibitor of CYP3A4 in the last 14 days; or
8. B12 deficiency not managed with intramuscular supplementation; or
9. Uncontrolled chronic diarrhea; or
10. Cirrhosis, or chronic active hepatitis; or
11. Pre-existent neuromuscular disease or persistent serum CK level > 3 times the upper limit of normal as measured within the past 60 days and determined to be non-transient through repeat testing; or
12. Patient with any of the following within the past 60 days:

    * white blood cell count < 3.0 X 109/L; or
    * platelet count <110 X 109/L; or
    * ALT or AST > 3 times the upper limit of normal (ULN); or
    * total bilirubin > 2 times ULN and not due to Gilbert syndrome.
13. Patient is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Dose tolerance | Up to 17 weeks
  Proportion of participants who permanently discontinue colchicine at either the 0.3 mg daily dose or 0.6 mg daily dose (to estimate the proportion who would discontinue the study drug at the 0.6 mg daily dose without titration).
Early discontinuations | Up to 17 weeks
  Proportion of participants who permanently discontinue colchicine at the 0.3 mg daily dose.

SECONDARY OUTCOMES:
Reason for drug discontinuation | Up to 17 weeks
  To determine the reasons for temporary and permanent discontinuations of colchicine at the 0.3 mg and 0.6 mg daily doses.
Drug adherence | Up to 17 weeks
  To determine degree of adherence to colchicine at the 0.3 mg and 0.6 mg daily doses.
Major Side Effects | Up to 17 weeks
  To determine the risk of major side effects of colchicine at the 0.3 mg and 0.6 mg daily doses.

OTHER OUTCOMES:
Colchicine Concentration | Up to 17 weeks
  To determine serum concentrations of colchicine achieved at the study doses.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Walsh, MD, PhD, Principal Investigator — McMaster University
Locations (3):
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: No